CLINICAL TRIAL: NCT06477315
Title: Mid- and Long-term Evaluation of the Results of Patients Undergoing Spinal Cord Stimulation With Microfractures + BST CarGel in the Treatment of Patellofemoral Chondral Lesions of the Knee
Acronym: CARGEL-LT
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: CARGEL-LT
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Chondral Lesion of the Knee; Patellofemoral Disorder
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- post surgery patients
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — telephone surveys

SUMMARY:
The study consists of 3 phases (Identification of eligible patients, follow-up by telephone or telemedicine platform and the collection of study-specific clinical data of enrolled patients):

* Identification by trained medical personnel of subjects who meet the study inclusion criteria.
* Once the patient's Informed Consent has been obtained, the study-specific questionnaires will be submitted.
* Clinical score data will be collected from the questionnaires conducted at mid- and long-term follow-up of patients enrolled in the study. The data collected during the long-term follow-up will be used to evaluate the time course of the results obtained after treatment of osteochondral lesions of the patellar cartilage by spinal cord stimulation with microfractures

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged between 18 and 75 years;
* BMI up to 30 kg/m2;
* Patients without subsequent surgery on the patellofemoral cartilage of the knee undergoing treatment;
* Ability and consent of patients to actively participate in the rehabilitation protocol and clinical and radiological follow-up;
* Signature of informed consent
* availability
* Competent patients

Exclusion Criteria:

* Patients no longer available;
* Patients who do not agree to undergo assessment;
* Deceased patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing treatment of osteochondral lesions of patellar cartilage by spinal cord stimulation with microfractures + BST CarGel
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee | baseline (post surgery)
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathologies. The questionnaire examines 3 categories: symptoms, sports activity and knee function. According to this questionnaire, a score between 0 and 100 can be obtained, whereby a high score is associated with a high level of function and minor pain symptoms. A score of 100 is in fact interpreted as a condition in which there are neither limitations in conducting activities of daily living nor symptoms.
Knee Injury and Osteoarthritis Outcome Score | baseline (post surgery)
  The complete questionnaire consists of five subscales and covers: pain (9 items), symptoms (7 items of which two concern stiffness), functions and activities of daily living (17 items) physical function, sports and leisure activities (5 items) and quality of life in relation to the knee (4 items). All items of the relevant subscales have the same response mode, use a 5-point Likert scale and each question is assigned a score from 0 to 4, where 0 indicates "no difficulty" and 4 "severe difficulty".) Score range 0-100 for each subscale.
EuroQol visual analogue scale | baseline (post surgery)
  It is a visual analogue scale that has a range of scores between 0 (worst imaginable health condition) and 100 (best imaginable health condition).
Tegner Score | baseline (post surgery)
  allows one to estimate the motor activity level of a subject with a score between 0 and 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports, such as football at national or international level. This score is the one most commonly used to define the motor activity level of patients with knee disorders.
(EuroQoL) Current Health Assessment | baseline (post surgery)
  valuable tool for measuring a patient's quality of life
Patient Acceptable Symptom State | baseline (post surgery)
  Valuable tool for assessing patient satisfaction in view of their current degree of pain, function and daily activity
Final assessment of treatment | baseline (post surgery)
  The patient should indicate satisfaction and the relative degree of satisfaction with the treatment after a minimum of 5 years after the infiltrative treatment.
failure question | baseline (post surgery)
  the patient should indicate whether and when a new infiltrative or surgical treatment was performed. Questions will also be asked about possible complications and re-interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Strauss EJ, Galos DK. The evaluation and management of cartilage lesions affecting the patellofemoral joint. Curr Rev Musculoskelet Med. 2013 Jun;6(2):141-9. doi: 10.1007/s12178-013-9157-z. PMID 23392780
- [Result] Duncan RC, Hay EM, Saklatvala J, Croft PR. Prevalence of radiographic osteoarthritis--it all depends on your point of view. Rheumatology (Oxford). 2006 Jun;45(6):757-60. doi: 10.1093/rheumatology/kei270. Epub 2006 Jan 17. PMID 16418199